CLINICAL TRIAL: NCT01110473
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetics of ABT-348 as Monotherapy and in Combination With Azacitidine in Subjects With Advanced Hematologic Malignancies
Brief Title: ABT-348 as Monotherapy and in Combination With Azacitidine to Treat Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-943
Record Dates: First submitted 2010-03-26; First posted 2010-04-26 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2013-11

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; B-cell Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Myelodysplasia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts | interventions — ilorasertib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Monotherapy, once daily (Experimental)
  Interventions: Drug: ABT-348
- Monotherapy, twice daily (Experimental)
  Interventions: Drug: ABT-348
- Combination with Azacitidine (Experimental)
  Interventions: Drug: ABT-348; Drug: ABT-348 and azacitidine
- IV monotherapy, once daily (Experimental)
  Interventions: Drug: ABT-348

INTERVENTIONS:
Drug: ABT-348 — An oral dose of ABT-348, once daily on Day 1, Day 8, and Day 15 of each 28 day cycle.
  Arms: Combination with Azacitidine; Monotherapy, once daily
Drug: ABT-348 — An oral dose of ABT-348, twice daily on Day 1, Day 8, and Day 15 of each 28 day cycle
  Arms: Monotherapy, twice daily
Drug: ABT-348 and azacitidine — An oral dose of ABT-348 on Day 1, Day 8, and Day 15 of each 28 day cycle. An IV or injection of azacitidine on Days 1-7 of each 28 day cycle.
  Arms: Combination with Azacitidine
Drug: ABT-348 — An intravenous dose of ABT-348, once daily on Day 1, Day 8, and Day 15 of each 28 day cycle.
  Arms: IV monotherapy, once daily

SUMMARY:
The purpose of this study is to determine the safety, pharmacokinetics and maximum tolerated dose of ABT-348 as monotherapy and when given in combination with azacitidine.

DETAILED DESCRIPTION:
The primary objectives of this study are to determine safety and pharmacokinetics of ABT-348 as monotherapy and when given in combination with azacitidine. The secondary objectives are to determine the maximum tolerated dose and recommended Phase 2 dose of ABT-348 when administered as monotherapy and when given in combination with azacitidine in subjects with advanced hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of one of the following (Arms A, B and D):

   * Relapsed or refractory acute myelogenous leukemia (AML), untreated AML in subjects who are > 60 years of age and do not have favorable cytogenetics (i.e., lack t(8,21) or inv(16)/t(16,16) or acute lymphoblastic leukemia (ALL) in subjects who have failed or are unsuitable for standard therapy.
   * Chronic myelogenous leukemia (CML) subjects that have not responded or relapsed on imatinib and failed second line Tyrosine Kinase Inhibitor (TKI) therapy and are not a candidate for allogeneic bone marrow transplant.
   * B-cell chronic lymphocytic leukemia (CLL) subjects that have not responded or relapsed on fludarabine or in the opinion of the Principal Investigator are unsuitable for fludarabine therapy and have not responded to or relapsed on alkylating therapy.
   * Myelodysplasia (MDS) including chronic myelomonocytic leukemia (CMML) subjects with International Prognostic Scoring System (IPSS) risk categories of Intermediate-2 (INT-2) or High risk, or any myelodysplasia with symptomatic anemia resistant to erythropoietin, immunosuppressant, or DNA methyltransferase inhibitor therapy (e.g., azacitidine/decitabine).

     1a. Histological or cytological confirmation of one of the following (Arm C):
   * Relapsed or refractory AML, untreated AML in subjects who are > 60 years of age and do not have favorable cytogenetics (i.e., lack t(8,21).
   * Untreated MDS including CMML with IPSS risk categories of INT-2 or High risk or with more than 10% blasts in the bone marrow, or any myelodysplasia with symptomatic anemia resistant to erythropoietin, or immunosuppressant, or subject has no response after four cycles of DNA methyltransferase inhibitor therapy or subject has progressed on DNA methyltransferase inhibitor therapy.
2. Eastern Cooperative Oncology Group Status of 0-2
3. Hematologic function for subjects with CLL and CML demonstrated by hemoglobin > 9 g/dL, platelets > 100,000/µL, ANC > 1500/mm3
4. Serum creatinine value of ≤ 1.8 times the upper limit of normal (ULN) and either an estimated creatinine clearance value as determined by the Cockcroft-Gault formula or based on a 24 hour urine collection creatinine clearance value of ≥ 50 mL/min
5. Adequate liver function as demonstrated by serum bilirubin < 2 x ULN and AST and ALT < 2.5 x ULN
6. QTc interval < 500 msec
7. Left Ventricular Ejection Fraction > 50%
8. Women of child-bearing potential and men must agree to use adequate contraception prior to the study entry, for the duration of study participation and up to 3 months following completion of therapy.
9. Capable of understanding and complying with parameters as outlined in the protocol and able to sign informed consent, approved by an Institutional Review Board (IRB) prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. Subject has known active CNS involvement. The subject has untreated brain or meningeal metastases.
2. ALL or AML subject has received acute anti-cancer therapy within 14 days prior to Study Day 1
3. CML, CLL or myelodysplasia (MDS) subjects has received acute anti-cancer therapy within 28 days or biologic therapy within 6 weeks prior to Study Day 1. Per Investigator discretion, hydroxyurea may be used anytime during the study. Tyrosine kinase inhibitors may not be administered 7 days prior to Study Day 1.
4. Subjects with poorly controlled diabetes mellitus
5. Subject has unresolved toxicities from prior anti-cancer therapy, grade 2 or higher clinically significant toxicity (excluding alopecia)
6. Subject has had major surgery within 28 days prior to Study Day 1
7. Subject currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure > 90 mmHg or systolic blood pressure > 140 mmHg
8. Subject has proteinuria grade > 1
9. Subject is unable to swallow or absorb oral tablets normally
10. Subject is receiving therapeutic anticoagulation therapy. Low-dose anticoagulation (e.g., low-dose heparin or warfarin) for catheter prophylaxis will be allowed
11. Subject has infection with HIV, Hepatitis B, or Hepatitis C
12. Female subjects who are pregnant or breast feeding
13. Any medical condition which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities
14. Clinically significant uncontrolled condition(s)
15. Subjects in Arm C who have advanced malignant hepatic tumors
16. Subjects in Arm C who have hypersensitivity to azacitidine or mannitol
17. Subjects have received CYP3A inhibitors or inducers within 7 days prior to the first dose of study drug.
18. Subjects enrolled in Arm D who have hypersensitivity to drugs formulated with polyethoxylated castor oil (Cremophor).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety profile (adverse events by toxicity grade and relationship to study drug, serious adverse events, adverse events leading to discontinuation and relevant clinical laboratory abnormalities) of ABT-348 as monotherapy or in combination | At each treatment visit
Study the pharmacokinetic interaction (plasma concentrations and pharmacokinetic parameter values) of ABT-348 as monotherapy and in combination | At study visits

SECONDARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RPTD) of ABT-348 when administered as a monotherapy and in combination in subjects with advanced hematologic malignancies | At each treatment visit

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gordon, MD, Study Director — AbbVie
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 59324, Scottsdale, Arizona
  - Site Reference ID/Investigator# 26523, Atlanta, Georgia
  - Site Reference ID/Investigator# 26522, Houston, Texas

REFERENCES:
- [Result] Garcia-Manero G, Tibes R, Kadia T, Kantarjian H, Arellano M, Knight EA, Xiong H, Qin Q, Munasinghe W, Roberts-Rapp L, Ansell P, Albert DH, Oliver B, McKee MD, Ricker JL, Khoury HJ. Phase 1 dose escalation trial of ilorasertib, a dual Aurora/VEGF receptor kinase inhibitor, in patients with hematologic malignancies. Invest New Drugs. 2015 Aug;33(4):870-80. doi: 10.1007/s10637-015-0242-6. Epub 2015 May 2. PMID 25933833